CLINICAL TRIAL: NCT02985476
Title: Electronic Linkage for Inflammatory Bowel Disease to Deliver Joint Access to Health Reports
Acronym: ELIJAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phedra Dodds (Other)
Collaborators: Swansea University (Other); The Health Foundation (Other)
Responsible Party: Sponsor-Investigator, Phedra Dodds, Consultant Nurse, Swansea University
Organization: Swansea University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 40189
Record Dates: First submitted 2016-09-13; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Electronic health records; Health records personal
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional (Active Comparator): Care as usual plus 8 weekly ELIJAH health reports shared with the participant and General Practitioner for 6 months i.e.: My history, My plan, My Update delivered via post or by email (dependant on participant preference) in addition to care as usual.
  Interventions: Other: Health reports
- Observational (No Intervention): Care as usual dictated by disease pathway of diagnosed inflammatory bowel disease i.e.; access to out-patient and in-patient hospital based care and community health resources via General Practitioner.

INTERVENTIONS:
Other: Health reports — Participants were sent 3 sets of individualised, educationally enriched health reports about their diagnosed inflammatory bowel disease history, care plan and updates on their recent health status, results or encounters with health care services.
  Arms: Interventional

SUMMARY:
This study evaluated the extent to which a shared health record facilitated better communication, increase individual responsibility for health care and reduce demand for health resources.

The study made individualised reports available to patients and General Practitioners and gave much more detail about participants chronic disease and treatments, and evaluated its effectiveness in a randomised controlled feasibility trial.

One third of patients received care as usual, two thirds of patients received the intervention.

DETAILED DESCRIPTION:
Chronic illness is a major cause of health problems. Self-management programmes can improve care and reduce healthcare resource use, but rely on well educated patients who are able to take responsibility for their care, have effective communication with health care providers, and easy access to appropriately triaged services.

This study utilised Inflammatory Bowel Disease as an exemplar of chronic disease management.

To inform the intervention the investigators held a focus group with patients who told the investigators about their concerns relating to education, care planning and communication about their condition. The participants expressed a preference for individualised information about their care, and plans of what to do if symptoms increase.

The investigators departmental electronic patient record (GeneCIS), was extended to provide personalised, educationally enriched information to each participant about their Inflammatory Bowel Disease. The investigators customised GeneCIS to develop output reports i.e.: "My History", "My plan" and "My Update", that attach specific educational information to the detailed, structured clinical data held on the system, and shared this with participants and their General Practitioner.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Inflammatory Bowel Disease, specifically Ulcerative Colitis or Crohn's Disease.
2. Aged 18 to 90 years.
3. Under the care of Consultant Gastroenterologists.
4. Patient registered with collaborating General Practitioner practice.

Exclusion Criteria:

a. Participants who are unable to comprehend the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety: Number of participants with adverse events as assessed by access to the primary and secondary care participant data and collated via the ELIJAH Adverse Event screening form. | 6 months
  The number of participants with adverse events leading to a hospital admission or otherwise, threatening the health and well being of participating patients and reported to a health professional graded according to causality and seriousness of event. Access to General Practitioner and secondary care hospital based data for the participant in paper and electronic form will provide details of relevant primary and secondary care attendances, acute admissions and outpatient appointments.

SECONDARY OUTCOMES:
Effectiveness: The cost of National Health Services resources used by participants in primary and secondary care. | 6 months
  The indirect costs of participant use of National Health services across primary and secondary care including General Practitioner visits, in-patient stays, operations, outpatient visits, investigations, Accident and Emergency attendances, open access service use and medication use will be compared. A direct cost of the intervention i.e.: the time taken by the clinician to formulate the elements of the ELIJAH intervention will be assessed. Both indirect and direct costs will be formulated via a comparrison of the PSSRU and National Schedule of reference Costs.
Patient- centeredness: Participant satisfaction with disease related care provided as assessed by Inflammatory Bowel Disease Service Satisfaction Questionnaire (ISSQ, derived from the GESQ). | 6 months
  Participant satisfaction of the care they receive.
Patient- centeredness: Participant satisfaction with disease related care provided as assessed by EQ5D. | 6 months
  Participant satisfaction of the care they receive.
Timeliness: The average elapsed time between the onset of a new inflammatory bowel disease related issue needing a healthcare intervention for a participant, and the start of that care. | 6 months
  Recognition of participants noting increased symptoms , the time of reporting symptoms and response time of health professionals to respond.
Equity: Whether the social status of participants affects the size of differences in the other four outcome criteria. | 6 months
  The number of participants designated by deprivation score (more or less deprived) using analysis of postcodes.

CONTACTS AND LOCATIONS:
Overall Officials: John G Williams, MSc, Principal Investigator — Professor of Health Services Research
Locations (1):
- Neath Port Talbot Hospital, Port Talbot, West Glamorgan, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data for the primary and secondary outcomes data will be made available upon completion of reporting of the trial.

REFERENCES:
- [Background] Travis SP, Stange EF, Lemann M, Oresland T, Bemelman WA, Chowers Y, Colombel JF, D'Haens G, Ghosh S, Marteau P, Kruis W, Mortensen NJ, Penninckx F, Gassull M; European Crohn's and Colitis Organisation (ECCO). European evidence-based Consensus on the management of ulcerative colitis: Current management. J Crohns Colitis. 2008 Mar;2(1):24-62. doi: 10.1016/j.crohns.2007.11.002. Epub 2008 Jan 18. No abstract available. PMID 21172195
- [Background] Stange EF, Travis SP, Vermeire S, Reinisch W, Geboes K, Barakauskiene A, Feakins R, Flejou JF, Herfarth H, Hommes DW, Kupcinskas L, Lakatos PL, Mantzaris GJ, Schreiber S, Villanacci V, Warren BF; European Crohn's and Colitis Organisation (ECCO). European evidence-based Consensus on the diagnosis and management of ulcerative colitis: Definitions and diagnosis. J Crohns Colitis. 2008 Mar;2(1):1-23. doi: 10.1016/j.crohns.2007.11.001. Epub 2008 Jan 18. No abstract available. PMID 21172194
- [Background] Williams JG, Cheung WY, Russell IT, Cohen DR, Longo M, Lervy B. Open access follow up for inflammatory bowel disease: pragmatic randomised trial and cost effectiveness study. BMJ. 2000 Feb 26;320(7234):544-8. doi: 10.1136/bmj.320.7234.544. PMID 10688560
- [Background] Robinson A, Thompson DG, Wilkin D, Roberts C; Northwest Gastrointestinal Research Group. Guided self-management and patient-directed follow-up of ulcerative colitis: a randomised trial. Lancet. 2001 Sep 22;358(9286):976-81. doi: 10.1016/S0140-6736(01)06105-0. PMID 11583752
- [Background] Osman LM, Abdalla MI, Beattie JA, Ross SJ, Russell IT, Friend JA, Legge JS, Douglas JG. Reducing hospital admission through computer supported education for asthma patients. Grampian Asthma Study of Integrated Care (GRASSIC). BMJ. 1994 Feb 26;308(6928):568-71. doi: 10.1136/bmj.308.6928.568. PMID 8093148
- [Background] Politi P, Bodini P, Mortilla MG, Beltrami M, Fornaciari G, Formisano D, Munkholm P, Riis L, Wolters F, Hoie O, Katsanos K, O'Morain C, Shuhaibar M, Lalli P, De Falco M, Pereira S, Freitas J, Odes S, Stockbrugger RW; European Collaborative Study Group on Inflammatory Bowel Disease. Communication of information to patients with inflammatory bowel disease: A European Collaborative Study in a multinational prospective inception cohort. J Crohns Colitis. 2008 Sep;2(3):226-32. doi: 10.1016/j.crohns.2008.01.007. Epub 2008 May 16. PMID 21172215
- [Background] Richardson G, Bloor K, Williams J, Russell I, Durai D, Cheung WY, Farrin A, Coulton S. Cost effectiveness of nurse delivered endoscopy: findings from randomised multi-institution nurse endoscopy trial (MINuET). BMJ. 2009 Feb 10;338:b270. doi: 10.1136/bmj.b270. PMID 19208715